CLINICAL TRIAL: NCT02404311
Title: A Phase 1-2 Randomized, Double-blind, Placebo-controlled Clinical Trial of Clade C ALVAC-HIV (vCP2438) and Bivalent Subtype C gp120/MF59® in HIV-uninfected Adults at Low Risk of HIV Infection
Brief Title: A Safety and Immune Response Study of 2 Experimental HIV Vaccines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); Bill and Melinda Gates Foundation (Other); Medical Research Council (Other Government); Sanofi Pasteur, a Sanofi Company (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 100
Record Dates: First submitted 2015-03-17; First posted 2015-03-31 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2020-07

CONDITIONS: HIV Infection
Keywords: HIV; AIDS; Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — AIDSVAX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part A, Group 1: Vaccine (Active Comparator): ALVAC-HIV at months 0 and 1, and ALVAC-HIV + bivalent subtype C gp120/MF59 at months 3, 6, and 12
  Interventions: Biological: ALVAC-HIV; Biological: Bivalent Subtype C gp120/MF59®
- Part A, Group 2: Placebo (Placebo Comparator): Placebo for ALVAC-HIV at months 0 and 1, and placebo for ALVAC-HIV + placebo for bivalent subtype C gp120/MF59 at months 3, 6, and 12
  Interventions: Biological: ALVAC-HIV (vCP2438) Placebo; Biological: Bivalent gp120/MF59® Placebo
- Part B, Group 1a: Vaccine (Active Comparator): Participants originally in Part A Group 1 (Vaccine) receive ALVAC-HIV + bivalent subtype C gp120/MF59 at month 30
  Interventions: Biological: ALVAC-HIV; Biological: Bivalent Subtype C gp120/MF59®
- Part B, Group 1b: Vaccine + Placebo (Active Comparator): Participants originally in Part A Group 1 (Vaccine) receive placebo for ALVAC-HIV + bivalent subtype C gp120/MF59 at month 30
  Interventions: Biological: Bivalent Subtype C gp120/MF59®; Biological: ALVAC-HIV (vCP2438) Placebo
- Part B, Group 2: Placebo (Placebo Comparator): Participants originally in Part A Group 2 (Placebo) receive placebo for ALVAC-HIV + placebo for bivalent subtype C gp120/MF59 at month 30
  Interventions: Biological: ALVAC-HIV (vCP2438) Placebo; Biological: Bivalent gp120/MF59® Placebo

INTERVENTIONS:
Biological: ALVAC-HIV — a lyophilized vaccine for injection at a viral titer ≥ 1 × 10E6 cell culture infectious dose (CCID)50 and < 1 × 10E8 CCID50 (nominal dose of 10E7 CCID50) and is reconstituted with 1mL of sterile sodium chloride solution (NaCl 0.4%) for intramuscular (IM) injection as a single dose.
  Arms: Part A, Group 1: Vaccine; Part B, Group 1a: Vaccine
Biological: Bivalent Subtype C gp120/MF59® — 2 recombinant monomeric proteins, each at a dose of 100 mcg, mixed with MF59® adjuvant (an oil-in-water emulsion) delivered as a 0.5 mL IM injection
  Arms: Part A, Group 1: Vaccine; Part B, Group 1a: Vaccine; Part B, Group 1b: Vaccine + Placebo
Biological: ALVAC-HIV (vCP2438) Placebo — a sterile, lyophilized product that consists of a mixture of virus stabilizer, and freeze drying medium and is reconstituted with 1mL of sterile sodium chloride solution (NaCl 0.4%) for injection as a single dose IM
  Arms: Part A, Group 2: Placebo; Part B, Group 1b: Vaccine + Placebo; Part B, Group 2: Placebo
Biological: Bivalent gp120/MF59® Placebo — Sodium chloride for injection, 0,9% delivered as a 0.5 mL IM injection
  Arms: Part A, Group 2: Placebo; Part B, Group 2: Placebo

SUMMARY:
The HIV Vaccine Trials Network (HVTN) is doing a study to test a new HIV vaccine combination. HIV is the virus that causes AIDS.

252 people are taking part in this study at multiple sites. The US National Institutes of Health (NIH) is paying for the study.

The investigators are doing this study to answer several questions.

* Are the study vaccines safe to give to people?
* Are people able to take the study vaccines without becoming too uncomfortable?
* How do people's immune systems respond to the study vaccines? (Your immune system protects you from disease.)

DETAILED DESCRIPTION:
The HIV Vaccine Trials Network (HVTN) is doing a study to test a new HIV vaccine combination. HIV is the virus that causes AIDS. The investigators are doing this study to answer several questions:

* Are the study vaccines safe to give to people?
* Are people able to take the study vaccines without becoming too uncomfortable?
* How do people's immune systems respond to the study vaccines? (Your immune system protects you from disease.)

The study uses 2 different vaccines: ALVAC-HIV (vCP2438) and bivalent gp120/MF59. These are experimental HIV vaccines -- the investigators do not know whether the vaccines will be safe to use in people, or whether they will work to prevent HIV infection. These vaccines are used only in research studies.

The ALVAC vaccine is made out of canarypox virus, which infects birds but cannot grow in human cells. This virus has small bits of man-made DNA inserted into it. DNA is a natural substance found in all living things, including people and some viruses. The canarypox virus helps get the DNA into the body's cells. The DNA then tells those cells to make small amounts of proteins that look like some of the ones found in HIV.

A study in South Africa, HVTN 097, gave a similar ALVAC vaccine to about 80 participants. So far, no one has had serious health problems.

The Protein vaccine has man-made pieces of a protein found on the outside of HIV. These protein pieces are mixed with an adjuvant called MF59. An adjuvant is something added to the vaccine to help the immune system respond better. MF59 has been included with other vaccines that have been given to over 50,000 people in clinical trials without causing any serious health problems.

This combination of study vaccines has not been given to people before. However, similar ALVAC and protein vaccines have been given to more than 10,000 people in clinical trials without causing any serious health problems. Also, over 300 people have received a similar combination of ALVAC and protein vaccines with the MF59 adjuvant in clinical trials without having any serious health problems.

The study is in 2 parts, Part A and Part B. Part B continues the study in order to learn how well boosting the study vaccines improves immune responses. 252 people took part in Part A of this study at multiple sites. Those who continue to meet eligibility requirements are invited to continue in Part B.

The US National Institutes of Health (NIH) is paying for the study. For people who continue to Part B, the study requires about 23 clinic visits in 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 40 years
* Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection (per Low Risk Guidelines for South African sites) and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Hemoglobin ≥ 11.0 g/dL for volunteers who were born female, ≥ 13.0 g/dL for volunteers who were born male
* WBC = 3,300 to 12,000 cells/mm3
* Total lymphocyte count ≥ 800 cells/mm3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets = 125,000 to 550,000/mm3
* Chemistry panel: ALT, AST, and ALP < 1.25 times the institutional upper limit of normal; creatinine ≤ institutional upper limit of normal.
* Negative HIV-1 and -2 blood test: Sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).
* Volunteers who were born female: negative urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination or negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test within 24 hours prior to initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy with bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception for participants in South Africa is defined as using 2 methods, including the following:
  * Condoms (male or female), or
  * Diaphragm or cervical cap,

PLUS 1 of the following methods:

* Intrauterine device (IUD),
* Hormonal contraception (in accordance with Republic of South Africa: National Contraception Clinical Guidelines),
* Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy); or
* Any other contraceptive method approved by the HVTN 100 PSRT
* Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
* Or be sexually abstinent.

  * Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) ≥ 40; or BMI ≥ 35 with 2 or more of the following: systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any study that includes HIV testing during the planned duration of the HVTN 100 study
* Pregnant, breastfeeding, or lactating
* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 100 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the South Africa Medicines Control Council (MCC). For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 100 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 100 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded from participation: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components such as eggs, egg products, or neomycin, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency
* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild or moderate, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses high dose inhaled corticosteroids, or
  * In the past year has either of the following:
  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, MBChB, DTMH, DCH, FCP(SA), PhD, Study Chair — HIV Vaccine Trials Network
Locations (5):
- South Africa (5):
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Isipingo CRS, Durban, KwaZulu-Natal
  - Emavundleni Desmond Tutu HIV Centre CRS, Cape Town, Western Cape
  - Aurum Institute for Health Research, Klerksdorp
  - Perinatal HIV Research Unit, Soweto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Naicker V, Laher F, Bekker LG, Seaton KE, Allen M, De Rosa S, Yates NL, Mkhize NN, Saunders K, Heptinstall J, Malahleha M, Mngadi K, Daniels B, Innes C, Yu C, Modise T, Bekker V, Grunenberg N, Furch B, Miner MD, Phogat S, Diazgranados CA, Gurunathan S, Koutsoukos M, Van Der Meeren O, Roxby AC, Ferrari G, Morris L, Montefiori D, McElrath MJ, Tomaras GD, Moodie Z. Safety and immunogenicity after a 30-month boost of a subtype C ALVAC-HIV (vCP2438) vaccine prime plus bivalent subtype C gp120/MF59 vaccine boost (HVTN 100): A phase 1-2 randomized double-blind placebo-controlled trial. PLOS Glob Public Health. 2024 Sep 20;4(9):e0003319. doi: 10.1371/journal.pgph.0003319. eCollection 2024. PMID 39302924
- [Derived] Hanass-Hancock J, Carpenter B, Reddy T, Nzuza A, Gaffoor Z, Goga A, Andrasik M. Participants' characteristics and motivations to screen for HIV vaccine and monoclonal antibody trials in KwaZulu-Natal, South Africa. Trials. 2021 Dec 11;22(1):897. doi: 10.1186/s13063-021-05792-7. PMID 34895272
- [Derived] Laher F, Moodie Z, Cohen KW, Grunenberg N, Bekker LG, Allen M, Frahm N, Yates NL, Morris L, Malahleha M, Mngadi K, Daniels B, Innes C, Saunders K, Grant S, Yu C, Gilbert PB, Phogat S, DiazGranados CA, Koutsoukos M, Van Der Meeren O, Bentley C, Mkhize NN, Pensiero MN, Mehra VL, Kublin JG, Corey L, Montefiori DC, Gray GE, McElrath MJ, Tomaras GD. Safety and immune responses after a 12-month booster in healthy HIV-uninfected adults in HVTN 100 in South Africa: A randomized double-blind placebo-controlled trial of ALVAC-HIV (vCP2438) and bivalent subtype C gp120/MF59 vaccines. PLoS Med. 2020 Feb 24;17(2):e1003038. doi: 10.1371/journal.pmed.1003038. eCollection 2020 Feb. PMID 32092060
- [Derived] Zhao LP, Fiore-Gartland A, Carpp LN, Cohen KW, Rouphael N, Fleurs L, Dintwe O, Zhao M, Moodie Z, Fong Y, Garrett N, Huang Y, Innes C, Janes HE, Lazarus E, Michael NL, Nitayaphan S, Pitisuttithum P, Rerks-Ngarm S, Robb ML, De Rosa SC, Corey L, Gray GE, Seaton KE, Yates NL, McElrath MJ, Frahm N, Tomaras GD, Gilbert PB. Landscapes of binding antibody and T-cell responses to pox-protein HIV vaccines in Thais and South Africans. PLoS One. 2020 Jan 30;15(1):e0226803. doi: 10.1371/journal.pone.0226803. eCollection 2020. PMID 31999736
- [Derived] Bekker LG, Moodie Z, Grunenberg N, Laher F, Tomaras GD, Cohen KW, Allen M, Malahleha M, Mngadi K, Daniels B, Innes C, Bentley C, Frahm N, Morris DE, Morris L, Mkhize NN, Montefiori DC, Sarzotti-Kelsoe M, Grant S, Yu C, Mehra VL, Pensiero MN, Phogat S, DiazGranados CA, Barnett SW, Kanesa-Thasan N, Koutsoukos M, Michael NL, Robb ML, Kublin JG, Gilbert PB, Corey L, Gray GE, McElrath MJ; HVTN 100 Protocol Team. Subtype C ALVAC-HIV and bivalent subtype C gp120/MF59 HIV-1 vaccine in low-risk, HIV-uninfected, South African adults: a phase 1/2 trial. Lancet HIV. 2018 Jul;5(7):e366-e378. doi: 10.1016/S2352-3018(18)30071-7. Epub 2018 Jun 18. PMID 29898870

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who received all vaccinations in Part A and completed Part A as scheduled were eligible for the Part B extension study. N=63 vaccination recipients in Part A (Group 1) were re-randomized to Part B Group 1a or 1b with a 1:1 ratio, while N=7 placebo recipients from Part A (Group 2) re-enrolled to receive placebo injections in Part B.
Groups:
- Part A, Group 1: Vaccine: Participants receive ALVAC-HIV (vCP2438) injections at months 0 and 1, and ALVAC-HIV (vCP2438) + bivalent subtype C gp120/MF59® injections at months 3, 6, and 12.
- Part A, Group 2: Placebo: Participants receive placebo for ALVAC-HIV (vCP2438) at months 0 and 1, and placebo for ALVAC-HIV (vCP2438) + placebo for bivalent subtype C gp120/MF59® injections at months 3, 6, and 12.
- Part B, Group 1a: Vaccine: Participants originally in Part A Group 1 receive ALVAC-HIV (vCP2438) + bivalent subtype C gp120/MF59® (vCP2438) injections at month 30.
- Part B, Group 1b: Vaccine + Placebo: Participants originally in Part A Group 1 receive placebo for ALVAC-HIV (vCP2438) + active bivalent subtype C gp120/MF59® at month 30.
- Part B, Group 2: Placebo: Participants originally in Part A Group 2 (Placebo) receive placebo for ALVAC-HIV (vCP2438) + placebo for bivalent subtype C gp120/MF59® at month 30.
Period: Part A: Month 0-18
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine + Placebo | Part B, Group 2: Placebo
Started | 210 | 42 | 0 | 0 | 0
Per Protocol | 185 | 37 | 0 | 0 | 0
Month 6.5 Immunogenicity Timepoint | 194 | 37 | 0 | 0 | 0
Month 12.5 Immunogenicity Timepoint | 186 | 33 | 0 | 0 | 0
Completed | 184 | 36 | 0 | 0 | 0
Not Completed | 26 | 6 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 0 | 0 | 0
Not completed — HIV Infection | 6 | 2 | 0 | 0 | 0
Not completed — Participant unable to adhere | 7 | 0 | 0 | 0 | 0
Period: Part B: Month 30-36
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine + Placebo | Part B, Group 2: Placebo
Started | 0 | 0 | 32 | 31 | 7
Month 30.5 Immunogenicity Timepoint | 0 | 0 | 28 | 30 | 6
Completed | 0 | 0 | 32 | 31 | 7
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A Only: Group 1 (Vaccine): Participants did not go on to Part B. In Part A, participants received ALVAC-HIV at months 0 and 1, and ALVAC-HIV + bivalent subtype C gp120/MF59 at months 3, 6, and 12
- Part A Only: Group 2 (Placebo): Participants did not go on to Part B. In Part A, participants received Placebo for ALVAC-HIV at months 0 and 1, and placebo for ALVAC-HIV + placebo for bivalent subtype C gp120/MF59 at months 3, 6, and 12
- Part A, Group 1 (Vaccine) + Part B, Group 1a (Vaccine): Participants completed Part A in Group 1 (Vaccine), joined Part B and were randomized to Group 1a (Vaccine): ALVAC-HIV + bivalent subtype C gp120/MF59 at month 30
- Part A, Group 1 (Vaccine) + Part B, Group 1b: Vaccine/Placeb: Participants completed Part A in Group 1 (Vaccine), joined Part B and were randomized to Group 1b (Vaccine/Placebo ): placebo for ALVAC-HIV + bivalent subtype C gp120/MF59 at month 30
- Part A, Group 2 (Placebo) + Part B, Group 2 (Placebo): Participants completed Part A in Group 2 (Placebo), joined Part B and received placebo for ALVAC-HIV + placebo for bivalent subtype C gp120/MF59 at month 30
- Total: Total of all reporting groups
Arm/Group | Part A Only: Group 1 (Vaccine) | Part A Only: Group 2 (Placebo) | Part A, Group 1 (Vaccine) + Part B, Group 1a (Vaccine) | Part A, Group 1 (Vaccine) + Part B, Group 1b: Vaccine/Placeb | Part A, Group 2 (Placebo) + Part B, Group 2 (Placebo) | Total
Number analyzed (Participants) | 147 | 35 | 32 | 31 | 7 | 252
Age, Continuous [Median (Full Range); unit: years] | 23 [18 to 40] | 23 [18 to 38] | 25 [19 to 38] | 23 [19 to 32] | 24 [19 to 39] | 23 [18 to 40]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 38 | 7 | 7 | 3 | 1 | 56
  21 - 30 years | 95 | 24 | 17 | 26 | 5 | 167
  31 - 40 years | 14 | 4 | 8 | 2 | 1 | 29
  41 - 50 years | 0 | 0 | 0 | 0 | 0 | 0
  Above 50 years | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 18 | 12 | 12 | 3 | 109
  Male | 83 | 17 | 20 | 19 | 4 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 147 | 35 | 32 | 31 | 7 | 252
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 143 | 34 | 31 | 31 | 7 | 246
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 3 | 1 | 1 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 147 | 35 | 32 | 31 | 7 | 252

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants Reporting Local Reactogenicity Signs and Symptoms During the Primary Vaccine Regimen
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017] The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 days after participants' last vaccination at Month 0,1,3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
Participants
  Pain: None | 42 | 26
  Pain: Mild | 126 | 16
  Pain: Moderate | 40 | 0
  Pain: Severe | 2 | 0
  Pain: Life Threatening | 0 | 0
  Tenderness: None | 69 | 34
  Tenderness: Mild | 114 | 8
  Tenderness: Moderate | 26 | 0
  Tenderness: Severe | 1 | 0
  Tenderness: Life Threatening | 0 | 0
  Pain and/or Tenderness: None | 35 | 26
  Pain and/or Tenderness: Mild | 131 | 16
  Pain and/or Tenderness: Moderate | 42 | 0
  Pain and/or Tenderness: Severe | 2 | 0
  Pain and/or Tenderness: Life Threatening | 0 | 0
  Erythema: None | 201 | 42
  Erythema: Mild | 6 | 0
  Erythema: Moderate | 2 | 0
  Erythema: Severe | 1 | 0
  Erythema: Life Threatening | 0 | 0
  Induration: None | 187 | 42
  Induration: Mild | 13 | 0
  Induration: Moderate | 9 | 0
  Induration: Severe | 1 | 0
  Induration: Life Threatening | 0 | 0
  Erythema and/or Induration: None | 185 | 42
  Erythema and/or Induration: Mild | 14 | 0
  Erythema and/or Induration: Moderate | 10 | 0
  Erythema and/or Induration: Severe | 1 | 0
  Erythema and/or Induration: Life Threatening | 0 | 0

2. Primary Outcome: Part A: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms During the Primary Vaccine Regimen
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Time Frame: Measured through 3 days after each vaccination at Month 0, 1, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
Participants
  Malaise and/or fatigue: None | 125 | 28
  Malaise and/or fatigue: Mild | 76 | 13
  Malaise and/or fatigue: Moderate | 9 | 1
  Malaise and/or fatigue: Severe | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0
  Myalgia: None | 132 | 34
  Myalgia: Mild | 60 | 7
  Myalgia: Moderate | 18 | 1
  Myalgia: Severe | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0
  Headache: None | 139 | 21
  Headache: Mild | 56 | 15
  Headache: Moderate | 15 | 6
  Headache: Severe | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0
  Nausea: None | 179 | 39
  Nausea: Mild | 29 | 3
  Nausea: Moderate | 2 | 0
  Nausea: Severe | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0
  Vomiting: None | 200 | 41
  Vomiting: Mild | 9 | 1
  Vomiting: Moderate | 1 | 0
  Vomiting: Severe | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0
  Chills: None | 195 | 40
  Chills: Mild | 14 | 2
  Chills: Moderate | 1 | 0
  Chills: Severe | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0
  Arthralgia: None | 151 | 33
  Arthralgia: Mild | 53 | 8
  Arthralgia: Moderate | 4 | 1
  Arthralgia: Severe | 2 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0
  Max. Systemic Symptoms: None | 68 | 16
  Max. Systemic Symptoms: Mild | 109 | 18
  Max. Systemic Symptoms: Moderate | 31 | 8
  Max. Systemic Symptoms: Severe | 2 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0
  Temperature: None | 195 | 41
  Temperature: Mild | 8 | 0
  Temperature: Moderate | 7 | 1
  Temperature: Severe | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity
Description: From the study termination form, early termination reasons associated with an AE or reactogenicity are tabulated by treatment arm
Time Frame: Measured through Month 18
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
Participants
  Termination due to AE/Reactogenicity | 4 | 2
  Other Reasons | 206 | 40

4. Primary Outcome: Part A: Number of Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: From the study product discontinuation form, study product administration reasons are tabulated by treatment arm
Time Frame: Measured through the Month 12 vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
Participants
  Clinical Event | 1 | 0
  Reactogenicity | 1 | 0
  Other Reasons | 19 | 3
  No Discontinuation | 189 | 39

5. Primary Outcome: Part A: Chemistry and Hematology Laboratory Results With Grade 1 or Higher
Description: Laboratory results are summarized by analyte and timepoint. Analytes and timepoint combinations with no grade 1 or higher results are not shown.
Time Frame: Measured during screening for part A, and 2 weeks after each vaccination at Month 0, 1, 3, 6, and 12
Population: The "overall number of participants analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, or they missed the scheduled visit, or they terminated participation in the study prior to the scheduled visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
Participants
  WBC (1000/cubic mm)-Screening | 0 | 0
  WBC (1000/cubic mm)-Day 14: number analyzed (Participants) | 207 | 41
  WBC (1000/cubic mm)-Day 14 | 0 | 0
  WBC (1000/cubic mm)-Day 42: number analyzed (Participants) | 202 | 40
  WBC (1000/cubic mm)-Day 42 | 0 | 0
  WBC (1000/cubic mm)-Day 98: number analyzed (Participants) | 198 | 39
  WBC (1000/cubic mm)-Day 98 | 0 | 0
  WBC (1000/cubic mm)-Day 182: number analyzed (Participants) | 195 | 37
  WBC (1000/cubic mm)-Day 182 | 0 | 0
  WBC (1000/cubic mm)-Day 378: number analyzed (Participants) | 187 | 36
  WBC (1000/cubic mm)-Day 378 | 0 | 0
  Neutrophils (1000/cubic mm)-Screening | 0 | 0
  Neutrophils (1000/cubic mm)-Day 14: number analyzed (Participants) | 207 | 41
  Neutrophils (1000/cubic mm)-Day 14 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 42: number analyzed (Participants) | 202 | 40
  Neutrophils (1000/cubic mm)-Day 42 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 98: number analyzed (Participants) | 198 | 39
  Neutrophils (1000/cubic mm)-Day 98 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 182: number analyzed (Participants) | 195 | 37
  Neutrophils (1000/cubic mm)-Day 182 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 378: number analyzed (Participants) | 187 | 36
  Neutrophils (1000/cubic mm)-Day 378 | 0 | 0
  Hemoglobin (g/dL)-Screening | 0 | 0
  Hemoglobin (g/dL)-Day 14: number analyzed (Participants) | 207 | 41
  Hemoglobin (g/dL)-Day 14 | 0 | 0
  Hemoglobin (g/dL)-Day 42: number analyzed (Participants) | 202 | 40
  Hemoglobin (g/dL)-Day 42 | 0 | 0
  Hemoglobin (g/dL)-Day 98: number analyzed (Participants) | 198 | 39
  Hemoglobin (g/dL)-Day 98 | 0 | 0
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 195 | 37
  Hemoglobin (g/dL)-Day 182 | 0 | 0
  Hemoglobin (g/dL)-Day 378: number analyzed (Participants) | 187 | 36
  Hemoglobin (g/dL)-Day 378 | 1 | 0
  Lymphocytes (1000/cubic mm)-Screening | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 14: number analyzed (Participants) | 207 | 41
  Lymphocytes (1000/cubic mm)-Day 14 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 42: number analyzed (Participants) | 202 | 40
  Lymphocytes (1000/cubic mm)-Day 42 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 98: number analyzed (Participants) | 198 | 39
  Lymphocytes (1000/cubic mm)-Day 98 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 182: number analyzed (Participants) | 195 | 37
  Lymphocytes (1000/cubic mm)-Day 182 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 378: number analyzed (Participants) | 187 | 36
  Lymphocytes (1000/cubic mm)-Day 378 | 0 | 0
  Platelets (1000/cubic mm)-Screening | 0 | 0
  Platelets (1000/cubic mm)-Day 14: number analyzed (Participants) | 207 | 41
  Platelets (1000/cubic mm)-Day 14 | 0 | 0
  Platelets (1000/cubic mm)-Day 42: number analyzed (Participants) | 201 | 40
  Platelets (1000/cubic mm)-Day 42 | 0 | 0
  Platelets (1000/cubic mm)-Day 98: number analyzed (Participants) | 198 | 39
  Platelets (1000/cubic mm)-Day 98 | 0 | 0
  Platelets (1000/cubic mm)-Day 182: number analyzed (Participants) | 194 | 37
  Platelets (1000/cubic mm)-Day 182 | 0 | 0
  Platelets (1000/cubic mm)-Day 378: number analyzed (Participants) | 187 | 36
  Platelets (1000/cubic mm)-Day 378 | 0 | 0
  ALT (SGPT) (U/L)-Screening | 0 | 0
  ALT (SGPT) (U/L)-Day 14: number analyzed (Participants) | 206 | 41
  ALT (SGPT) (U/L)-Day 14 | 0 | 0
  ALT (SGPT) (U/L)-Day 42: number analyzed (Participants) | 203 | 40
  ALT (SGPT) (U/L)-Day 42 | 1 | 0
  ALT (SGPT) (U/L)-Day 98: number analyzed (Participants) | 198 | 39
  ALT (SGPT) (U/L)-Day 98 | 1 | 0
  ALT (SGPT) (U/L)-Day 182: number analyzed (Participants) | 195 | 37
  ALT (SGPT) (U/L)-Day 182 | 0 | 0
  ALT (SGPT) (U/L)-Day 378: number analyzed (Participants) | 188 | 36
  ALT (SGPT) (U/L)-Day 378 | 1 | 0
  AST (U/L)-Screening | 0 | 0
  AST (U/L)-Day 14: number analyzed (Participants) | 207 | 41
  AST (U/L)-Day 14 | 0 | 0
  AST (U/L)-Day 42: number analyzed (Participants) | 203 | 40
  AST (U/L)-Day 42 | 2 | 0
  AST (U/L)-Day 98: number analyzed (Participants) | 198 | 39
  AST (U/L)-Day 98 | 0 | 0
  AST (U/L)-Day 182: number analyzed (Participants) | 195 | 37
  AST (U/L)-Day 182 | 0 | 0
  AST (U/L)-Day 378: number analyzed (Participants) | 188 | 36
  AST (U/L)-Day 378 | 1 | 0
  Alkaline Phosphatase (U/L)-Screening | 0 | 0
  Alkaline Phosphatase (U/L)-Day 14: number analyzed (Participants) | 207 | 41
  Alkaline Phosphatase (U/L)-Day 14 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 42: number analyzed (Participants) | 203 | 40
  Alkaline Phosphatase (U/L)-Day 42 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 98: number analyzed (Participants) | 198 | 39
  Alkaline Phosphatase (U/L)-Day 98 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 182: number analyzed (Participants) | 195 | 37
  Alkaline Phosphatase (U/L)-Day 182 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 378: number analyzed (Participants) | 188 | 36
  Alkaline Phosphatase (U/L)-Day 378 | 0 | 0
  Creatinine (g/dL)-Screening | 0 | 0
  Creatinine (g/dL)-Day 14: number analyzed (Participants) | 207 | 41
  Creatinine (g/dL)-Day 14 | 0 | 0
  Creatinine (g/dL)-Day 42: number analyzed (Participants) | 203 | 40
  Creatinine (g/dL)-Day 42 | 1 | 0
  Creatinine (g/dL)-Day 98: number analyzed (Participants) | 198 | 39
  Creatinine (g/dL)-Day 98 | 0 | 0
  Creatinine (g/dL)-Day 182: number analyzed (Participants) | 194 | 37
  Creatinine (g/dL)-Day 182 | 0 | 0
  Creatinine (g/dL)-Day 378: number analyzed (Participants) | 188 | 36
  Creatinine (g/dL)-Day 378 | 3 | 0

6. Primary Outcome: Part A Chemistry Laboratory Measures: Alkaline Phosphatase, AST, and ALT
Description: For each chemistry laboratory measure, summary statistics were presented by analyte and treatment group for the overall population.
Time Frame: Time Frame: Measured during screening for part A, and 2 weeks after each vaccination at Month 0, 1, 3, 6, and 12
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
U/L
  ALT (SGPT) (U/L)-Screening | 17 [13 to 24] | 19 [13 to 24]
  ALT (SGPT) (U/L)-Day 14: number analyzed (Participants) | 206 | 41
  ALT (SGPT) (U/L)-Day 14 | 17 [13 to 22] | 19 [14 to 22]
  ALT (SGPT) (U/L)-Day 42: number analyzed (Participants) | 203 | 40
  ALT (SGPT) (U/L)-Day 42 | 19 [14 to 28] | 21 [14.5 to 27]
  ALT (SGPT) (U/L)-Day 98: number analyzed (Participants) | 198 | 39
  ALT (SGPT) (U/L)-Day 98 | 18.5 [13 to 26] | 18 [14 to 22]
  ALT (SGPT) (U/L)-Day 182: number analyzed (Participants) | 195 | 37
  ALT (SGPT) (U/L)-Day 182 | 19 [13 to 25] | 19 [15 to 23]
  ALT (SGPT) (U/L)-Day 378: number analyzed (Participants) | 188 | 36
  ALT (SGPT) (U/L)-Day 378 | 20 [15 to 30] | 21 [17 to 27]
  AST (U/L)-Screening | 22 [19 to 26] | 22 [19 to 26]
  AST (U/L)-Day 14: number analyzed (Participants) | 207 | 41
  AST (U/L)-Day 14 | 22 [19 to 25] | 21 [18 to 24]
  AST (U/L)-Day 42: number analyzed (Participants) | 203 | 40
  AST (U/L)-Day 42 | 23 [19 to 29] | 23 [19 to 27.5]
  AST (U/L)-Day 98: number analyzed (Participants) | 198 | 39
  AST (U/L)-Day 98 | 23 [20 to 28] | 23 [21 to 27]
  AST (U/L)-Day 182: number analyzed (Participants) | 195 | 37
  AST (U/L)-Day 182 | 24 [21 to 29] | 25 [21 to 28]
  AST (U/L)-Day 378: number analyzed (Participants) | 188 | 36
  AST (U/L)-Day 378 | 24 [20 to 28.5] | 22.5 [20 to 26]
  Alkaline Phosphatase (U/L)-Screening | 71.5 [56 to 85] | 72.5 [57 to 87]
  Alkaline Phosphatase (U/L)-Day 14: number analyzed (Participants) | 207 | 41
  Alkaline Phosphatase (U/L)-Day 14 | 69 [57 to 83] | 71 [56 to 81]
  Alkaline Phosphatase (U/L)-Day 42: number analyzed (Participants) | 203 | 40
  Alkaline Phosphatase (U/L)-Day 42 | 70 [59 to 86] | 71 [58 to 87.5]
  Alkaline Phosphatase (U/L)-Day 98: number analyzed (Participants) | 198 | 39
  Alkaline Phosphatase (U/L)-Day 98 | 73 [60 to 87] | 74 [62 to 85]
  Alkaline Phosphatase (U/L)-Day 182: number analyzed (Participants) | 195 | 37
  Alkaline Phosphatase (U/L)-Day 182 | 69 [59 to 83] | 70 [59 to 85]
  Alkaline Phosphatase (U/L)-Day 378: number analyzed (Participants) | 188 | 36
  Alkaline Phosphatase (U/L)-Day 378 | 72 [60.5 to 87] | 74.5 [61.5 to 86.5]

7. Primary Outcome: Part A Chemistry Laboratory Measures: Hemoglobin, Creatinine
Description: as for outcome 6
Time Frame: Time Frame: Measured during screening for part A, and 2 weeks after each vaccination at Month 0, 1, 3, 6, and 12
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
g/dL
  Hemoglobin (g/dL)-Screening | 14.7 [13.6 to 15.7] | 14.4 [13.1 to 15.9]
  Hemoglobin (g/dL)-Day 14: number analyzed (Participants) | 207 | 41
  Hemoglobin (g/dL)-Day 14 | 14.1 [12.9 to 15.2] | 13.4 [12.3 to 15]
  Hemoglobin (g/dL)-Day 42: number analyzed (Participants) | 202 | 40
  Hemoglobin (g/dL)-Day 42 | 14.4 [13.3 to 15.6] | 13.75 [12.45 to 15.2]
  Hemoglobin (g/dL)-Day 98: number analyzed (Participants) | 198 | 39
  Hemoglobin (g/dL)-Day 98 | 14.3 [13.3 to 15.5] | 13.5 [12.7 to 15.5]
  Hemoglobin (g/dL)-Day 182: number analyzed (Participants) | 195 | 37
  Hemoglobin (g/dL)-Day 182 | 14.1 [12.9 to 15.2] | 13.9 [12.8 to 14.9]
  Hemoglobin (g/dL)-Day 378: number analyzed (Participants) | 187 | 36
  Hemoglobin (g/dL)-Day 378 | 13.9 [12.7 to 14.7] | 13.4 [12.35 to 15.35]
  Creatinine (g/dL)-Screening | 0.0007 [0.00063 to 0.00081] | 0.0007 [0.0006 to 0.0008]
  Creatinine (g/dL)-Day 14: number analyzed (Participants) | 207 | 41
  Creatinine (g/dL)-Day 14 | 0.00077 [0.00063 to 0.0009] | 0.0007 [0.00063 to 0.0008]
  Creatinine (g/dL)-Day 42: number analyzed (Participants) | 203 | 40
  Creatinine (g/dL)-Day 42 | 0.0007 [0.00068 to 0.00081] | 0.0007 [0.000605 to 0.000855]
  Creatinine (g/dL)-Day 98: number analyzed (Participants) | 198 | 39
  Creatinine (g/dL)-Day 98 | 0.00073 [0.00066 to 0.00081] | 0.00077 [0.0006 to 0.0009]
  Creatinine (g/dL)-Day 182: number analyzed (Participants) | 194 | 37
  Creatinine (g/dL)-Day 182 | 0.0008 [0.00069 to 0.0009] | 0.0007 [0.00062 to 0.0008]
  Creatinine (g/dL)-Day 378: number analyzed (Participants) | 188 | 36
  Creatinine (g/dL)-Day 378 | 0.0008 [0.0007 to 0.0009] | 0.0007 [0.000635 to 0.0008]

8. Primary Outcome: Part A Hematology Laboratory Measures: WBC, Platelets, Lymphocytes, Neutrophils
Description: as for outcome 6
Time Frame: Measured during screening for part A, and 2 weeks after each vaccination at Month 0, 1, 3, 6, and 12
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
thousand cells/cubic mm
  WBC (1000/cubic mm)-Screening | 6.135 [5.06 to 7.6] | 6.3 [5.5 to 7.7]
  WBC (1000/cubic mm)-Day 14: number analyzed (Participants) | 207 | 41
  WBC (1000/cubic mm)-Day 14 | 6 [4.84 to 7.29] | 5.9 [4.54 to 7.02]
  WBC (1000/cubic mm)-Day 42: number analyzed (Participants) | 202 | 40
  WBC (1000/cubic mm)-Day 42 | 5.87 [4.6 to 6.9] | 5.425 [4.395 to 7.1]
  WBC (1000/cubic mm)-Day 98: number analyzed (Participants) | 198 | 39
  WBC (1000/cubic mm)-Day 98 | 6.055 [4.76 to 7.32] | 5.9 [4.44 to 7.2]
  WBC (1000/cubic mm)-Day 182: number analyzed (Participants) | 195 | 37
  WBC (1000/cubic mm)-Day 182 | 5.67 [4.7 to 6.9] | 5.63 [4.1 to 6.71]
  WBC (1000/cubic mm)-Day 378: number analyzed (Participants) | 187 | 36
  WBC (1000/cubic mm)-Day 378 | 5.69 [4.72 to 7] | 5.815 [4.5 to 7.18]
  Neutrophils (1000/cubic mm)-Screening | 3.23 [2.38 to 4.419] | 3.265 [2.41 to 4.16]
  Neutrophils (1000/cubic mm)-Day 14: number analyzed (Participants) | 207 | 41
  Neutrophils (1000/cubic mm)-Day 14 | 3.18 [2.233 to 4.217] | 3.08 [1.987 to 4.107]
  Neutrophils (1000/cubic mm)-Day 42: number analyzed (Participants) | 202 | 40
  Neutrophils (1000/cubic mm)-Day 42 | 3.057 [2.159 to 4.02] | 2.9015 [1.7805 to 4.18]
  Neutrophils (1000/cubic mm)-Day 98: number analyzed (Participants) | 198 | 39
  Neutrophils (1000/cubic mm)-Day 98 | 3.284 [2.251 to 4.627] | 3.25 [2.302 to 3.99]
  Neutrophils (1000/cubic mm)-Day 182: number analyzed (Participants) | 195 | 37
  Neutrophils (1000/cubic mm)-Day 182 | 2.927 [2.219 to 4.09] | 2.629 [1.796 to 4.02]
  Neutrophils (1000/cubic mm)-Day 378: number analyzed (Participants) | 187 | 36
  Neutrophils (1000/cubic mm)-Day 378 | 3.08 [2.22 to 3.99] | 3.089 [1.802 to 4.1015]
  Lymphocytes (1000/cubic mm)-Screening | 2.182 [1.84 to 2.546] | 2.299 [1.947 to 2.66]
  Lymphocytes (1000/cubic mm)-Day 14: number analyzed (Participants) | 207 | 41
  Lymphocytes (1000/cubic mm)-Day 14 | 2.102 [1.731 to 2.434] | 2.064 [1.84 to 2.31]
  Lymphocytes (1000/cubic mm)-Day 42: number analyzed (Participants) | 202 | 40
  Lymphocytes (1000/cubic mm)-Day 42 | 2.0545 [1.663 to 2.39] | 2.031 [1.72 to 2.375]
  Lymphocytes (1000/cubic mm)-Day 98: number analyzed (Participants) | 198 | 39
  Lymphocytes (1000/cubic mm)-Day 98 | 1.9435 [1.657 to 2.35] | 2.02 [1.777 to 2.58]
  Lymphocytes (1000/cubic mm)-Day 182: number analyzed (Participants) | 195 | 37
  Lymphocytes (1000/cubic mm)-Day 182 | 2.004 [1.675 to 2.41] | 1.96 [1.77 to 2.25]
  Lymphocytes (1000/cubic mm)-Day 378: number analyzed (Participants) | 187 | 36
  Lymphocytes (1000/cubic mm)-Day 378 | 2 [1.62 to 2.38] | 1.975 [1.6885 to 2.315]
  Platelets (1000/cubic mm)-Screening | 250.5 [213 to 295] | 275 [233 to 308]
  Platelets (1000/cubic mm)-Day 14: number analyzed (Participants) | 207 | 41
  Platelets (1000/cubic mm)-Day 14 | 265 [222 to 313] | 272 [227 to 311]
  Platelets (1000/cubic mm)-Day 42: number analyzed (Participants) | 201 | 40
  Platelets (1000/cubic mm)-Day 42 | 267 [223 to 313] | 270 [229.5 to 300]
  Platelets (1000/cubic mm)-Day 98: number analyzed (Participants) | 198 | 39
  Platelets (1000/cubic mm)-Day 98 | 267 [224 to 309] | 276 [234 to 321]
  Platelets (1000/cubic mm)-Day 182: number analyzed (Participants) | 194 | 37
  Platelets (1000/cubic mm)-Day 182 | 259.5 [220 to 303] | 267 [237 to 294]
  Platelets (1000/cubic mm)-Day 378: number analyzed (Participants) | 187 | 36
  Platelets (1000/cubic mm)-Day 378 | 273 [233 to 318] | 264.5 [244 to 307.5]

9. Primary Outcome: Part A: Occurrence of IgG Ab Binding to gp120 Env Proteins Contained in the Vaccine (ZM96, TV1.C, 1086.C) After the Primary Vaccine Regimen, Measured by HIV-1 Multiplex Antibody Assay
Description: Serum HIV-1-specific IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. Samples from post-enrollment visits have positive responses if they meet three conditions: (1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of pre-vaccination net MFI), (2) net MFI values are greater than 3 times pre-vaccination net MFI, and (3) experimental antigen MFI values are greater than 3 times pre-vaccination MFI. Data are excluded if the blood draw date was outside the allowable window, a participant was HIV-infected, or the reference antigen exceeds 5000 MFI.
Time Frame: Measured at Month 6.5
Population: "Overall Number of Participants Analyzed" includes those with samples collected at the month 6.5 immunogenicity timepoint, who were HIV-uninfected and received the first 4 vaccinations. "Number Analyzed" shows the number of participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 185 | 37
Participants
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 185 | 36
  1086C_D7gp120.avi/293F | 185 | 0
  96ZM651.D11gp120.avi: number analyzed (Participants) | 185 | 36
  96ZM651.D11gp120.avi | 185 | 0
  TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 185 | 36
  TV1c8_D11gp120.avi/293F | 185 | 0

10. Primary Outcome: Part A: Level of IgG Ab Binding to gp120 Env Proteins Contained in the Vaccine (ZM96, TV1.C, 1086.C) After the Primary Vaccine Regimen, Measured by HIV-1 Multiplex Antibody Assay
Description: Serum HIV-1-specific IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. The measure unit fluorescence units are relative to assay background, not relative to the placebo arm. Background is used here rather than negative control stimulation, since the antigens are used as bead coating rather than stimulation.
Time Frame: Measured at Month 6.5
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 185 | 37
fluorescence unit relative to background
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 185 | 36
  1086C_D7gp120.avi/293F | 28359.5 [25888 to 30784.25] | 1 [1 to 1]
  96ZM651.D11gp120.avi: number analyzed (Participants) | 185 | 36
  96ZM651.D11gp120.avi | 2650 [1536 to 4868.5] | 1 [1 to 1]
  TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 185 | 36
  TV1c8_D11gp120.avi/293F | 12883.5 [6023.5 to 22540.75] | 1 [1 to 1]

11. Primary Outcome: Part A: Occurrence of IgG Binding Antibodies to 3 V1V2-scaffolded Env Proteins After the Primary Vaccine Regimen
Description: Measured by HIV-1 multiplex Ab assay: refer to earlier description for assay methods and analysis variable derivation. The number and percentage of participants with positive responses are summarized by antigen.
Time Frame: Measured at Month 6.5
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 185 | 37
Participants
  C.1086C_V1_V2 Tags: number analyzed (Participants) | 183 | 35
  C.1086C_V1_V2 Tags | 129 | 0
  gp70-96ZM651.02 V1v2: number analyzed (Participants) | 181 | 35
  gp70-96ZM651.02 V1v2 | 88 | 0
  gp70-TV1.21 V1V2: number analyzed (Participants) | 183 | 35
  gp70-TV1.21 V1V2 | 113 | 0

12. Primary Outcome: Part A: Level of IgG Binding Antibodies to 3 V1V2-scaffolded Env Proteins After the Primary Vaccine Regimen
Description: as for outcome 10
Time Frame: Measured at Month 6.5
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 185 | 37
fluorescence unit relative to background
  C.1086C_V1_V2 Tags: number analyzed (Participants) | 183 | 35
  C.1086C_V1_V2 Tags | 562 [98.5 to 2085.75] | 1 [1 to 2.5]
  gp70-96ZM651.02 V1v2: number analyzed (Participants) | 181 | 35
  gp70-96ZM651.02 V1v2 | 392.5 [48 to 1008] | 1 [1 to 138]
  gp70-TV1.21 V1V2: number analyzed (Participants) | 183 | 35
  gp70-TV1.21 V1V2 | 338.25 [37.25 to 1188.3] | 1 [1 to 1]

13. Primary Outcome: Part A: Occurrence of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine After the Primary Vaccine Regimen. Measured by Flow Cytometry.
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers after peptide stimulation minus % cells expressing markers after no stimulation. A contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). A one-sided Fisher's exact test is applied, testing if the number of cells positive for the marker is equal in the stimulated vs. unstimulated cells. A discrete Bonferroni adjustment is made over the peptide pools. Response is positive if p<=0.00001. Data are excluded if the blood draw date was outside the visit window, the participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high.
Time Frame: Measured at Month 6.5
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 185 | 37
Participants
  Any gp120: number analyzed (Participants) | 181 | 34
  Any gp120 | 120 | 1
  1086 gp120: number analyzed (Participants) | 181 | 34
  1086 gp120 | 82 | 1
  TV1 gp120: number analyzed (Participants) | 181 | 34
  TV1 gp120 | 112 | 1
  ZM96 gp120: number analyzed (Participants) | 181 | 34
  ZM96 gp120 | 102 | 0

14. Primary Outcome: Part A: Level of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine After the Primary Vaccine Regimen.
Description: Measured by flow cytometry ICS assay: refer to earlier description for assay methods and analysis variable derivation. Percentage of T-cells expressing cytokines are summarized for positive responders only.
Time Frame: Measured at Month 6.5
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 185 | 37
% CD4+ T-cells
  Any gp120: number analyzed (Participants) | 181 | 34
  Any gp120 | 0.11501130 [0.06637581 to 0.1965080] | 0.003579320 [-0.00316960 to 0.02699403]
  1086 gp120: number analyzed (Participants) | 181 | 34
  1086 gp120 | 0.06613413 [0.03475199 to 0.1374808] | -0.00296204 [-0.01473795 to 0.00669736]
  TV1 gp120: number analyzed (Participants) | 181 | 34
  TV1 gp120 | 0.09629575 [0.05269700 to 0.1701793] | -0.002244635 [-0.01399708 to 0.00818973]
  ZM96 gp120: number analyzed (Participants) | 181 | 34
  ZM96 gp120 | 0.0889934 [0.0443736 to 0.1742616] | -0.002505630 [-0.00943639 to 0.00967744]

15. Primary Outcome: Part B: Number of Participants Reporting Local Reactogenicity Signs and Symptoms in the Extension Study
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]. For each participant, the maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 days after the Month 30 vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Part B, Group 1b: Vaccine/Placebo: Participants originally in Part A Group 1 (Vaccine) receive placebo for ALVAC-HIV + bivalent subtype C gp120/MF59 at month 30
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
Participants
  Pain: None | 16 | 18 | 7
  Pain: Mild | 12 | 11 | 0
  Pain: Moderate | 4 | 2 | 0
  Pain: Severe | 0 | 0 | 0
  Pain: Life Threatening | 0 | 0 | 0
  Tenderness: None | 21 | 25 | 7
  Tenderness: Mild | 7 | 5 | 0
  Tenderness: Moderate | 4 | 1 | 0
  Tenderness: Severe | 0 | 0 | 0
  Tenderness: Life Threatening | 0 | 0 | 0
  Pain and/or Tenderness: None | 14 | 17 | 7
  Pain and/or Tenderness: Mild | 11 | 12 | 0
  Pain and/or Tenderness: Moderate | 7 | 2 | 0
  Pain and/or Tenderness: Severe | 0 | 0 | 0
  Pain and/or Tenderness: Life Threatening | 0 | 0 | 0
  Erythema: None | 28 | 27 | 7
  Erythema: Mild | 1 | 3 | 0
  Erythema: Moderate | 3 | 1 | 0
  Erythema: Severe | 0 | 0 | 0
  Erythema: Life Threatening | 0 | 0 | 0
  Induration: None | 28 | 25 | 7
  Induration: Mild | 1 | 4 | 0
  Induration: Moderate | 2 | 1 | 0
  Induration: Severe | 1 | 1 | 0
  Induration: Life Threatening | 0 | 0 | 0
  Erythema and/or Induration: None | 28 | 24 | 7
  Erythema and/or Induration: Mild | 0 | 4 | 0
  Erythema and/or Induration: Moderate | 3 | 2 | 0
  Erythema and/or Induration: Severe | 1 | 1 | 0
  Erythema and/or Induration: Life Threatening | 0 | 0 | 0

16. Primary Outcome: Part B: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms in the Extension Study
Description: as for outcome 15
Time Frame: Measured through 3 days after the Month 30 vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
Participants
  Malaise and/or fatigue: None | 21 | 24 | 7
  Malaise and/or fatigue: Mild | 9 | 7 | 0
  Malaise and/or fatigue: Moderate | 2 | 0 | 0
  Malaise and/or fatigue: Severe | 0 | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0
  Myalgia: None | 21 | 24 | 7
  Myalgia: Mild | 7 | 7 | 0
  Myalgia: Moderate | 4 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0
  Headache: None | 26 | 29 | 6
  Headache: Mild | 6 | 2 | 1
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0
  Nausea: None | 31 | 30 | 7
  Nausea: Mild | 1 | 1 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0
  Vomiting: None | 32 | 30 | 7
  Vomiting: Mild | 0 | 1 | 0
  Vomiting: Moderate | 0 | 0 | 0
  Vomiting: Severe | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0
  Chills: None | 28 | 29 | 7
  Chills: Mild | 4 | 2 | 0
  Chills: Moderate | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0
  Arthralgia: None | 25 | 28 | 7
  Arthralgia: Mild | 6 | 3 | 0
  Arthralgia: Moderate | 1 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0
  Max. Systemic Symptoms: None | 16 | 21 | 6
  Max. Systemic Symptoms: Mild | 11 | 10 | 1
  Max. Systemic Symptoms: Moderate | 5 | 0 | 0
  Max. Systemic Symptoms: Severe | 0 | 0 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0
  Temperature: None | 32 | 31 | 7
  Temperature: Mild | 0 | 0 | 0
  Temperature: Moderate | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0

17. Primary Outcome: Part B: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity
Description: From the study termination form, early termination reasons associated with an AE are tabulated by treatment arm
Time Frame: Measured through Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
Participants
  Termination not due to AE/Reactogenicity | 0 | 0 | 0
  Other reason | 32 | 31 | 7

18. Primary Outcome: Part B: Chemistry and Hematology Laboratory Results of Grade 1 or Higher
Description: as for outcome 5
Time Frame: Time Frame: Measured during screening for part B, and 2 weeks after vaccination at Month 30
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
Participants
  WBC (1000/cubic mm)-Part B Screening | 0 | 0 | 0
  WBC (1000/cubic mm)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  WBC (1000/cubic mm)-Day 924 | 0 | 0 | 0
  Neutrophils (1000/cubic mm)-Part B Screening | 0 | 0 | 0
  Neutrophils (1000/cubic mm)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Neutrophils (1000/cubic mm)-Day 924 | 0 | 0 | 0
  Hemoglobin (g/dL)-Part B Screening | 0 | 0 | 0
  Hemoglobin (g/dL)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Hemoglobin (g/dL)-Day 924 | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)-Part B Screening | 0 | 0 | 0
  Lymphocytes (1000/cubic mm)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Lymphocytes (1000/cubic mm)-Day 924 | 0 | 0 | 0
  Platelets (1000/cubic mm)-Part B Screening: number analyzed (Participants) | 31 | 31 | 7
  Platelets (1000/cubic mm)-Part B Screening | 0 | 0 | 0
  Platelets (1000/cubic mm)-Day 924: number analyzed (Participants) | 27 | 30 | 6
  Platelets (1000/cubic mm)-Day 924 | 0 | 0 | 0
  ALT (SGPT) (U/L)-Part B Screening | 0 | 0 | 0
  ALT (SGPT) (U/L)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  ALT (SGPT) (U/L)-Day 924 | 0 | 0 | 0
  AST (U/L)-Part B Screening | 0 | 0 | 0
  AST (U/L)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  AST (U/L)-Day 924 | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Part B Screening | 0 | 0 | 0
  Alkaline Phosphatase (U/L)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Alkaline Phosphatase (U/L)-Day 924 | 0 | 0 | 0
  Creatinine (g/dL)-Part B Screening | 1 | 2 | 0
  Creatinine (g/dL)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Creatinine (g/dL)-Day 924 | 1 | 6 | 1

19. Primary Outcome: Part B Chemistry Laboratory Measures: Alkaline Phosphatase, AST, and ALT
Description: as for outcome 6
Time Frame: Measured during screening for part B, and 2 weeks after vaccination at Month 30
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
U/L
  ALT (SGPT) (U/L)-Part B Screening | 17 [12 to 23] | 18 [16 to 21] | 20 [12 to 23]
  ALT (SGPT) (U/L)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  ALT (SGPT) (U/L)-Day 924 | 16 [13 to 22] | 15 [12 to 22] | 16.5 [14 to 29]
  AST (U/L)-Part B Screening | 22.5 [18.5 to 26] | 23 [19 to 26] | 20 [19 to 22]
  AST (U/L)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  AST (U/L)-Day 924 | 20.5 [19 to 26] | 21 [19 to 23] | 22 [16 to 24]
  Alkaline Phosphatase (U/L)-Part B Screening | 73 [59 to 88] | 74 [64 to 90] | 68 [62 to 86]
  Alkaline Phosphatase (U/L)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Alkaline Phosphatase (U/L)-Day 924 | 76.5 [64.5 to 92] | 69 [56 to 79] | 59.5 [58 to 79]

20. Primary Outcome: Part B Chemistry Laboratory Measures: Hemoglobin, Creatinine
Description: as for outcome 6
Time Frame: Measured during screening for part B, and 2 weeks after vaccination at Month 30
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
g/dL
  Hemoglobin (g/dL)-Part B Screening | 14.85 [13.75 to 15.7] | 14.6 [12.9 to 15.6] | 13.8 [11.9 to 15.3]
  Hemoglobin (g/dL)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Hemoglobin (g/dL)-Day 924 | 14.65 [13.45 to 15.1] | 13.965 [12.1 to 15.2] | 13.7 [11.7 to 14.9]
  Creatinine (g/dL)-Part B Screening | 0.00085 [0.0007 to 0.001] | 0.0007 [0.0007 to 0.0008] | 0.0007 [0.0006 to 0.0008]
  Creatinine (g/dL)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Creatinine (g/dL)-Day 924 | 0.0009 [0.00072 to 0.00095] | 0.0008 [0.00061 to 0.0009] | 0.00075 [0.00069 to 0.0008]

21. Primary Outcome: Part B Chemistry Laboratory Measures: WBC, Platelets, Lymphocytes, Neutrophils
Description: as for outcome 6
Time Frame: Measured during screening for part B, and 2 weeks after vaccination at Month 30
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
thousand cells/cubic mm
  WBC (1000/cubic mm)-Part B Screening | 6.4 [5.45 to 7.79] | 6.59 [4.66 to 8.03] | 7.1 [5 to 8.03]
  WBC (1000/cubic mm)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  WBC (1000/cubic mm)-Day 924 | 6.28 [5.285 to 8.295] | 6.355 [4.67 to 6.93] | 6.505 [5.76 to 7.73]
  Neutrophils (1000/cubic mm)-Part B Screening | 3.499 [2.847 to 4.741] | 3.41 [2.54 to 4.959] | 3.38 [2.331 to 4.826]
  Neutrophils (1000/cubic mm)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Neutrophils (1000/cubic mm)-Day 924 | 3.577 [2.7545 to 5.1055] | 3.7825 [2.309 to 4.133] | 3.031 [2.92 to 4.352]
  Lymphocytes (1000/cubic mm)-Part B Screening | 2.2295 [1.859 to 2.5305] | 1.941 [1.682 to 2.583] | 2.559 [2.425 to 3.01]
  Lymphocytes (1000/cubic mm)-Day 924: number analyzed (Participants) | 28 | 30 | 6
  Lymphocytes (1000/cubic mm)-Day 924 | 2.031 [1.742 to 2.3985] | 1.9295 [1.666 to 2.093] | 2.541 [2.334 to 2.72]
  Platelets (1000/cubic mm)-Part B Screening: number analyzed (Participants) | 31 | 31 | 7
  Platelets (1000/cubic mm)-Part B Screening | 264 [225 to 291] | 256 [213 to 294] | 311 [265 to 343]
  Platelets (1000/cubic mm)-Day 924: number analyzed (Participants) | 27 | 30 | 6
  Platelets (1000/cubic mm)-Day 924 | 279 [240 to 317] | 248.5 [211 to 297] | 281.5 [277 to 297]

22. Primary Outcome: Part B: Occurrence of IgG Binding Antibodies to 3 V1V2-scaffolded Env Proteins in the Extension Study
Description: as for outcome 11
Time Frame: Measured at Month 30.5
Population: "Overall Number of Participants Analyzed" includes those with samples collected at month 30.5, who were HIV-uninfected and received the all vaccinations. "Number Analyzed" counts participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 28 | 30 | 6
Participants
  C.1086C_V1_V2 Tags: number analyzed (Participants) | 26 | 30 | 6
  C.1086C_V1_V2 Tags | 19 | 23 | 0
  gp70-96ZM651.02 V1v2: number analyzed (Participants) | 26 | 30 | 6
  gp70-96ZM651.02 V1v2 | 14 | 15 | 0
  gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 21 | 27 | 6
  gp70-TV1.GSKvacV1V2/293F | 15 | 18 | 0

23. Primary Outcome: Part B: Level of IgG Binding Antibodies to 3 V1V2-scaffolded Env Proteins in the Extension Study
Description: as for outcome 10
Time Frame: Measured at Month 30.5
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 28 | 30 | 6
fluorescence unit relative to background
  C.1086C_V1_V2 Tags: number analyzed (Participants) | 26 | 30 | 6
  C.1086C_V1_V2 Tags | 527.375 [156.25 to 1506.5] | 562.25 [171.25 to 2866.75] | 1 [1 to 1]
  gp70-96ZM651.02 V1v2: number analyzed (Participants) | 26 | 30 | 6
  gp70-96ZM651.02 V1v2 | 858.125 [159.75 to 17625.5] | 1015.625 [183.5 to 2618.5] | 1 [1 to 133.5]
  gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 21 | 27 | 6
  gp70-TV1.GSKvacV1V2/293F | 924.75 [304 to 6457.5] | 1537 [154.75 to 11308] | 1 [1 to 4.75]

24. Primary Outcome: Part B: Occurrence of IgG Ab Binding to gp120 Env Proteins Contained in the Vaccine (ZM96, TV1.C, 1086.C) in the Extension Study
Description: as for outcome 11
Time Frame: Measured at Month 30.5
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 28 | 30 | 6
Participants
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 26 | 30 | 6
  1086C_D7gp120.avi/293F | 26 | 30 | 0
  96ZM651.D11gp120.avi: number analyzed (Participants) | 26 | 30 | 6
  96ZM651.D11gp120.avi | 25 | 29 | 0
  TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 26 | 30 | 6
  TV1c8_D11gp120.avi/293F | 26 | 30 | 0

25. Primary Outcome: Part B: Level of IgG Ab Binding to gp120 Env Proteins Contained in the Vaccine (ZM96, TV1.C, 1086.C) in the Extension Study
Description: as for outcome 10
Time Frame: Measured at Month 30.5
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 28 | 30 | 6
fluorescence unit relative to background
  1086C_D7gp120.avi/293F: number analyzed (Participants) | 26 | 30 | 6
  1086C_D7gp120.avi/293F | 31063.875 [30695.25 to 31272] | 30887.75 [30415 to 31428.75] | 1 [1 to 1]
  96ZM651.D11gp120.avi: number analyzed (Participants) | 26 | 30 | 6
  96ZM651.D11gp120.avi | 30006.875 [29070.75 to 30465.25] | 30137.5 [28980 to 30938.25] | 1 [1 to 12.25]
  TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 26 | 30 | 6
  TV1c8_D11gp120.avi/293F | 30864.875 [30308 to 31304.75] | 30674.125 [30076.5 to 31240.25] | 1 [1 to 5.75]

26. Primary Outcome: Part B: Occurrence of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine in the Extension Study
Description: Measured by flow cytometry ICS assay: refer to earlier description for assay methods and analysis variable derivation. The number and percentage of participants with positive responses are summarized by peptide pool.
Time Frame: Measured at Month 30.5
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 28 | 30 | 6
Participants
  Any gp120: number analyzed (Participants) | 26 | 28 | 5
  Any gp120 | 25 | 26 | 0
  1086 gp120: number analyzed (Participants) | 26 | 28 | 5
  1086 gp120 | 22 | 23 | 0
  TV1 gp120: number analyzed (Participants) | 26 | 28 | 5
  TV1 gp120 | 24 | 25 | 0
  ZM96 gp120: number analyzed (Participants) | 26 | 28 | 5
  ZM96 gp120 | 23 | 22 | 0

27. Primary Outcome: Part B: Level of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine in the Extension Study
Description: as for outcome 14
Time Frame: Measured at Month 30.5
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: % of CD4+ T-cells
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 28 | 30 | 6
% of CD4+ T-cells
  Any gp120: number analyzed (Participants) | 26 | 28 | 5
  Any gp120 | 0.284956245 [0.11146075 to 0.38500129] | 0.18676016 [0.121813505 to 0.261912375] | 0.00889506 [0 to 0.0335174]
  1086 gp120: number analyzed (Participants) | 26 | 28 | 5
  1086 gp120 | 0.1299094 [0.06802766 to 0.27495601] | 0.11812899 [0.076206435 to 0.17014021] | -0.00507644 [-0.00912041 to -0.00408307]
  TV1 gp120: number analyzed (Participants) | 26 | 28 | 5
  TV1 gp120 | 0.23924445 [0.10696857 to 0.35719109] | 0.180244495 [0.086940765 to 0.242827475] | 0.00889506 [-0.01525722 to 0.00990069]
  ZM96 gp120: number analyzed (Participants) | 26 | 28 | 5
  ZM96 gp120 | 0.25434725 [0.10973632 to 0.33505092] | 0.13517637 [0.068628665 to 0.18483264] | -0.00325229 [-0.00701159 to -0.00203876]

28. Secondary Outcome: Part A: Frequency of Severe Local Reactogenicity Signs and Symptoms, Through the Fifth Vaccination
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 days after each vaccination at Month 0, 1, 3, 6, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
Participants
  Pain: None | 37 | 24
  Pain: Mild | 120 | 17
  Pain: Moderate | 50 | 1
  Pain: Severe | 3 | 0
  Pain: Life Threatening | 0 | 0
  Tenderness: None | 60 | 33
  Tenderness: Mild | 114 | 8
  Tenderness: Moderate | 35 | 1
  Tenderness: Severe | 1 | 0
  Tenderness: Life Threatening | 0 | 0
  Pain and/or Tenderness: None | 30 | 24
  Pain and/or Tenderness: Mild | 123 | 17
  Pain and/or Tenderness: Moderate | 54 | 1
  Pain and/or Tenderness: Severe | 3 | 0
  Pain and/or Tenderness: Life Threatening | 0 | 0
  Erythema: None | 196 | 42
  Erythema: Mild | 8 | 0
  Erythema: Moderate | 3 | 0
  Erythema: Severe | 3 | 0
  Erythema: Life Threatening | 0 | 0
  Induration: None | 178 | 42
  Induration: Mild | 17 | 0
  Induration: Moderate | 12 | 0
  Induration: Severe | 3 | 0
  Induration: Life Threatening | 0 | 0
  Erythema and/or Induration: None | 176 | 42
  Erythema and/or Induration: Mild | 17 | 0
  Erythema and/or Induration: Moderate | 14 | 0
  Erythema and/or Induration: Severe | 3 | 0
  Erythema and/or Induration: Life Threatening | 0 | 0

29. Secondary Outcome: Part A: Frequency of Severe Systemic Reactogenicity Signs and Symptoms, Through the Fifth Vaccination
Description: as for outcome 28
Time Frame: Measured through 3 days after each vaccination at Month 0, 1, 3, 6, and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo
Number analyzed (Participants) | 210 | 42
Participants
  Malaise and/or fatigue: None | 121 | 26
  Malaise and/or fatigue: Mild | 74 | 14
  Malaise and/or fatigue: Moderate | 15 | 1
  Malaise and/or fatigue: Severe | 0 | 1
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0
  Myalgia: None | 124 | 34
  Myalgia: Mild | 64 | 7
  Myalgia: Moderate | 22 | 1
  Myalgia: Severe | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0
  Headache: None | 130 | 19
  Headache: Mild | 62 | 17
  Headache: Moderate | 17 | 6
  Headache: Severe | 1 | 0
  Headache: Potentially Life-threatening | 0 | 0
  Nausea: None | 174 | 38
  Nausea: Mild | 34 | 4
  Nausea: Moderate | 2 | 0
  Nausea: Severe | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0
  Vomiting: None | 200 | 41
  Vomiting: Mild | 9 | 1
  Vomiting: Moderate | 1 | 0
  Vomiting: Severe | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0
  Chills: None | 187 | 40
  Chills: Mild | 21 | 2
  Chills: Moderate | 2 | 0
  Chills: Severe | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0
  Arthralgia: None | 143 | 33
  Arthralgia: Mild | 57 | 8
  Arthralgia: Moderate | 8 | 1
  Arthralgia: Severe | 2 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0
  Max. Systemic Symptoms: None | 63 | 14
  Max. Systemic Symptoms: Mild | 104 | 19
  Max. Systemic Symptoms: Moderate | 40 | 8
  Max. Systemic Symptoms: Severe | 3 | 1
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0
  Temperature: None | 192 | 41
  Temperature: Mild | 11 | 0
  Temperature: Moderate | 7 | 1
  Temperature: Severe | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0

30. Secondary Outcome: Part A: Compare the Occurrence of IgG Ab Binding to gp120 Env Proteins Contained in the Vaccine (ZM96, TV1.C, 1086.C) After the Fourth Versus the Fifth Vaccination
Description: as for outcome 9
Time Frame: Measured at Month 6.5 and 12.5
Population: The durability cohort was randomly selected from those in the month 6.5 cohort with samples collected at month 12.5. Selection was stratified by gender to match the overall protocol. "Overall Number of Participants Analyzed" represents the durability cohort. "Number Analyzed" counts participants with data meeting assay-specific quality criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine
Number analyzed (Participants) | 65
Participants
  1086C_D7gp120.avi/293F (Month 6.5) | 64
  1086C_D7gp120.avi/293F (Month 12.5) | 64
  96ZM651.D11gp120.avi (Month 6.5) | 59
  96ZM651.D11gp120.avi (Month 12.5) | 59
  TV1c8_D11gp120.avi/293F (Month 6.5) | 64
  TV1c8_D11gp120.avi/293F (Month 12.5) | 64
Statistical Analysis 1: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to 1086C_D7gp120.avi/293F after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 1.0000, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = -0.015 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 2: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to 96ZM651.D11gp120.avi after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 1.0000, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = -0.015 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 3: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to TV1c8_D11gp120.avi/293F after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 1.0000, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = -0.015 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)

31. Secondary Outcome: Part A: Compare the Level of IgG Ab Binding to gp120 Env Proteins Contained in the Vaccine (ZM96, TV1.C, 1086.C) After the Fourth Versus the Fifth Vaccination
Description: Serum HIV-1-specific IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. The measure unit fluorescence units are relative to assay background, not relative to the placebo arm. Background is used here rather than negative control stimulation, since the antigens are used as bead coating rather than stimulation. Comparisons were performed among positive responders only (positivity criteria is described in Outcome 30).
Time Frame: Measured at Month 6.5 and 12.5
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Part A, Group 1: Vaccine
Number analyzed (Participants) | 65
fluorescence unit relative to background
  1086C_D7gp120.avi/293F (Month 6.5) | 29317.375 [28375.25 to 29980.25]
  1086C_D7gp120.avi/293F (Month 12.5) | 31407.349999 [30676.474999 to 31978.475001]
  96ZM651.D11gp120.avi (Month 6.5) | 26437.25 [24669 to 28770.5]
  96ZM651.D11gp120.avi (Month 12.5) | 31378.5 [30576.5 to 31901.5]
  TV1c8_D11gp120.avi/293F (Month 6.5) | 28365.625 [27214.375 to 29583.25]
  TV1c8_D11gp120.avi/293F (Month 12.5) | 31425.5 [30760.475006 to 31893.375]
Statistical Analysis 1: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to 1086C_D7gp120.avi/293F after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p < .0001, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 0.914 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 2: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to 96ZM651.D11gp120.avi after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p < .0001, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 0.945 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 3: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to TV1c8_D11gp120.avi/293F after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p < .0001, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 0.895 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)

32. Secondary Outcome: Part A: Compare the Occurrence of IgG Binding Antibodies to 3 V1V2-scaffolded Env Proteins After the Fourth Versus the Fifth Vaccination
Description: as for outcome 9
Time Frame: Measured at Month 6.5 and 12.5
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine
Number analyzed (Participants) | 65
Participants
  C.1086C_V1_V2 Tags (Month 6.5) | 49
  C.1086C_V1_V2 Tags (Month 12.5) | 57
  gp70-96ZM651.02 V1v2 (Month 6.5) | 29
  gp70-96ZM651.02 V1v2 (Month 12.5) | 44
  gp70-TV1.GSKvacV1V2/293F (Month 6.5): number analyzed (Participants) | 57
  gp70-TV1.GSKvacV1V2/293F (Month 6.5) | 36
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 57
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 50
Statistical Analysis 1: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to C.1086C_V1_V2 Tags after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.0215, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = 0 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 2: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to gp70-96ZM651.02 V1v2 after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.0003, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = 0 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 3: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to gp70-TV1.GSKvacV1V2/293F after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.0010, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = 0.228 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)

33. Secondary Outcome: Part A: Compare the Level of IgG Binding Antibodies to 3 V1V2-scaffolded Env Proteins After the Fourth Versus the Fifth Vaccination
Description: Serum HIV-1-specific IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI less than 1 is set to 1. The measure unit fluorescence units are relative to assay background, not relative to the placebo arm. Background is used here rather than negative control stimulation, since the antigens are used as bead coating rather than stimulation. Comparisons were performed among positive responders only (positivity criteria is described in Outcome 32).
Time Frame: Measured at Month 6.5 and 12.5
Population: as for outcome 30
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Part A, Group 1: Vaccine
Number analyzed (Participants) | 65
fluorescence unit relative to background
  C.1086C_V1_V2 Tags (Month 6.5) | 1281.5 [662.75 to 2252]
  C.1086C_V1_V2 Tags (Month 12.5) | 2938.5 [1141.699997 to 6677.999806]
  gp70-96ZM651.02 V1v2 (Month 6.5) | 1747.5 [871.75 to 3196.25]
  gp70-96ZM651.02 V1v2 (Month 12.5) | 3821.75 [1544.4000245 to 9955.8500005]
  gp70-TV1.GSKvacV1V2/293F (Month 6.5): number analyzed (Participants) | 57
  gp70-TV1.GSKvacV1V2/293F (Month 6.5) | 3082.625 [1198.375 to 8855]
  gp70-TV1.GSKvacV1V2/293F (Month 12.5): number analyzed (Participants) | 57
  gp70-TV1.GSKvacV1V2/293F (Month 12.5) | 4207.8499015 [1341.5 to 13130.5]
Statistical Analysis 1: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to C.1086C_V1_V2 Tags after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p < .0001, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 0 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 2: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to gp70-96ZM651.02 V1v2 after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p < .0001, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 0 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 3: Comparison: Part A, Group 1: Vaccine; IgG Ab binding to gp70-TV1.GSKvacV1V2/293F after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.0002, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 6.099 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)

34. Secondary Outcome: Part A: Compare the Occurrence of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine After the Fourth Versus the Fifth Vaccinations
Description: as for outcome 13
Time Frame: Measured at Month 6.5 and 12.5
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Group 1: Vaccine
Number analyzed (Participants) | 56
Participants
  1086 gp120 (Month 6.5) | 24
  1086 gp120 (Month 12.5) | 23
  TV1 gp120 (Month 6.5) | 32
  TV1 gp120 (Month 12.5) | 31
  ZM96 gp120 (Month 6.5) | 30
  ZM96 gp120 (Month 12.5) | 34
Statistical Analysis 1: Comparison: Part A, Group 1: Vaccine; CD4+ T Cell Responses to 1086 gp120 after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 1.0000, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = 0.018 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 2: Comparison: Part A, Group 1: Vaccine; CD4+ T Cell Responses to TV1 gp120 after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.6698, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = 0.036 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 3: Comparison: Part A, Group 1: Vaccine; CD4+ T Cell Responses to ZM96 gp120 after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.1435, McNemar — The threshold for statistical significance was p = 0.05; Proportion Difference (Net) = 0.125 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)

35. Secondary Outcome: Part A: Compare the Level of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine After the Fourth Versus the Fifth Vaccinations
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing markers after peptide stimulation minus % cells expressing markers after no stimulation. A contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). A one-sided Fisher's exact test is applied, testing if the number of cells positive for the marker is equal in the stimulated vs. unstimulated cells. A discrete Bonferroni adjustment is made over the peptide pools. Response is positive if p<=0.00001. Data are excluded if the blood draw date was outside the visit window, the participant was HIV-infected, PBMC viability or T-cell count were low, or negative control was high. Comparisons were performed among positive responders only.
Time Frame: Measured at Month 6.5 and 12.5
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Part A, Group 1: Vaccine
Number analyzed (Participants) | 56
% CD4+ T-cells
  1086 gp120 (Month 6.5) | 0.17577251 [0.116401835 to 0.27437614]
  1086 gp120 (Month 12.5) | 0.14932756 [0.11886426 to 0.34311697]
  TV1 gp120 (Month 6.5) | 0.158423055 [0.12192562 to 0.354710545]
  TV1 gp120 (Month 12.5) | 0.22183561 [0.13385739 to 0.33774746]
  ZM96 gp120 (Month 6.5) | 0.17436147 [0.1468941 to 0.36994411]
  ZM96 gp120 (Month 12.5) | 0.203201925 [0.14269436 to 0.4014336]
Statistical Analysis 1: Comparison: Part A, Group 1: Vaccine; CD4+ T Cell Responses to 1086 gp120 after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.9661, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 0.965 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 2: Comparison: Part A, Group 1: Vaccine; CD4+ T Cell Responses to TV1 gp120 after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.8593, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 1.118 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)
Statistical Analysis 3: Comparison: Part A, Group 1: Vaccine; CD4+ T Cell Responses to ZM96 gp120 after the fourth (month 6.5) versus the fifth vaccination (month 12.5); Test type: Other; p = 0.4396, Wilcoxon Signed-Rank — The threshold for statistical significance was p = 0.05; Geometric Mean difference (Net) = 1.138 — Difference = Month 12.5 (5th vaccination) - Month 6.5 (4th vaccination)

36. Secondary Outcome: Part B: Occurrence of IgG Ab Binding to gp120 Env Proteins Contained in the Vaccine (ZM96, TV1.C, 1086.C) in the Extension Study, at 6 Months After the Month 30 Vaccination
Description: as for outcome 9
Time Frame: Measured at Month 30 and 36
Population: "Overall Number of Participants Analyzed" represents Part B participants. "Number Analyzed" counts participants with data meeting assay-specific quality criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
Participants
  1086C_D7gp120.avi/293F (Month 30): number analyzed (Participants) | 31 | 31 | 7
  1086C_D7gp120.avi/293F (Month 30) | 31 | 30 | 0
  1086C_D7gp120.avi/293F (Month 36): number analyzed (Participants) | 31 | 30 | 7
  1086C_D7gp120.avi/293F (Month 36) | 31 | 30 | 0
  96ZM651.D11gp120.avi (Month 30): number analyzed (Participants) | 31 | 31 | 7
  96ZM651.D11gp120.avi (Month 30) | 2 | 2 | 0
  96ZM651.D11gp120.avi (Month 36): number analyzed (Participants) | 31 | 30 | 7
  96ZM651.D11gp120.avi (Month 36) | 24 | 25 | 0
  TV1c8_D11gp120.avi/293F (Month 30): number analyzed (Participants) | 31 | 31 | 7
  TV1c8_D11gp120.avi/293F (Month 30) | 27 | 30 | 0
  TV1c8_D11gp120.avi/293F (Month 36): number analyzed (Participants) | 31 | 30 | 7
  TV1c8_D11gp120.avi/293F (Month 36) | 31 | 30 | 0

37. Secondary Outcome: Part B: Level of IgG Ab Binding to gp120 Env Proteins Contained in the Vaccine (ZM96, TV1.C, 1086.C) in the Extension Study, at 6 Months After the Month 30 Vaccination
Description: as for outcome 10
Time Frame: Measured at Month 30 and 36
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
fluorescence unit relative to background
  1086C_D7gp120.avi/293F (Month 30): number analyzed (Participants) | 31 | 31 | 7
  1086C_D7gp120.avi/293F (Month 30) | 6664 [2265.25 to 10900.5] | 4415 [2585.75 to 7880] | 1 [1 to 1]
  1086C_D7gp120.avi/293F (Month 36): number analyzed (Participants) | 31 | 30 | 7
  1086C_D7gp120.avi/293F (Month 36) | 25399 [21608.25 to 30932.25] | 24763.625 [18642.25 to 27445] | 1 [1 to 1]
  96ZM651.D11gp120.avi (Month 30): number analyzed (Participants) | 31 | 31 | 7
  96ZM651.D11gp120.avi (Month 30) | 895.25 [301.25 to 1278.5] | 706.5 [424.25 to 1566] | 1 [1 to 10.75]
  96ZM651.D11gp120.avi (Month 36): number analyzed (Participants) | 31 | 30 | 7
  96ZM651.D11gp120.avi (Month 36) | 9750 [2871 to 22625] | 7324.75 [4300.5 to 16439.25] | 2.75 [1 to 12]
  TV1c8_D11gp120.avi/293F (Month 30): number analyzed (Participants) | 31 | 31 | 7
  TV1c8_D11gp120.avi/293F (Month 30) | 937 [328.75 to 2063] | 616.25 [273.75 to 1288.5] | 1 [1 to 73.5]
  TV1c8_D11gp120.avi/293F (Month 36): number analyzed (Participants) | 31 | 30 | 7
  TV1c8_D11gp120.avi/293F (Month 36) | 17175.5 [5443.25 to 30353.75] | 17192.375 [9493 to 23194.25] | 1 [1 to 84.25]

38. Secondary Outcome: Part B: Occurrence of IgG Binding Antibodies to 3 V1V2-scaffolded Env Proteins in the Extension Study, at 6 Months After the Month 30 Vaccination
Description: as for outcome 9
Time Frame: Measured at Month 30 and 36
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
Participants
  C.1086C_V1_V2 Tags (Month 30): number analyzed (Participants) | 31 | 31 | 7
  C.1086C_V1_V2 Tags (Month 30) | 7 | 6 | 0
  C.1086C_V1_V2 Tags (Month 36): number analyzed (Participants) | 31 | 30 | 7
  C.1086C_V1_V2 Tags (Month 36) | 9 | 12 | 1
  gp70-96ZM651.02 V1v2 (Month 30): number analyzed (Participants) | 31 | 31 | 7
  gp70-96ZM651.02 V1v2 (Month 30) | 2 | 1 | 0
  gp70-96ZM651.02 V1v2 (Month 36): number analyzed (Participants) | 31 | 30 | 7
  gp70-96ZM651.02 V1v2 (Month 36) | 7 | 3 | 1
  gp70-TV1.GSKvacV1V2/293F (Month 30): number analyzed (Participants) | 25 | 27 | 6
  gp70-TV1.GSKvacV1V2/293F (Month 30) | 0 | 2 | 0
  gp70-TV1.GSKvacV1V2/293F (Month 36): number analyzed (Participants) | 25 | 26 | 6
  gp70-TV1.GSKvacV1V2/293F (Month 36) | 4 | 4 | 0

39. Secondary Outcome: Part B: Level of IgG Binding Antibodies to 3 V1V2-scaffolded Env Proteins in the Extension Study, at 6 Months After the Month 30 Vaccination
Description: as for outcome 10
Time Frame: Measured at Month 30 and 36
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: fluorescence unit relative to background
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
fluorescence unit relative to background
  C.1086C_V1_V2 Tags (Month 30): number analyzed (Participants) | 31 | 31 | 7
  C.1086C_V1_V2 Tags (Month 30) | 13.5 [8.25 to 89.5] | 23 [4.75 to 92] | 2.75 [1 to 61.75]
  C.1086C_V1_V2 Tags (Month 36): number analyzed (Participants) | 31 | 30 | 7
  C.1086C_V1_V2 Tags (Month 36) | 47.25 [12.75 to 152] | 79.25 [18.25 to 322.75] | 4.75 [1.75 to 80]
  gp70-96ZM651.02 V1v2 (Month 30): number analyzed (Participants) | 31 | 31 | 7
  gp70-96ZM651.02 V1v2 (Month 30) | 1 [1 to 246] | 1 [1 to 51.25] | 1 [1 to 333.5]
  gp70-96ZM651.02 V1v2 (Month 36): number analyzed (Participants) | 31 | 30 | 7
  gp70-96ZM651.02 V1v2 (Month 36) | 19.75 [1 to 1438] | 35.375 [1 to 166] | 1 [1 to 654.75]
  gp70-TV1.GSKvacV1V2/293F (Month 30): number analyzed (Participants) | 25 | 27 | 6
  gp70-TV1.GSKvacV1V2/293F (Month 30) | 1 [1 to 46.5] | 1 [1 to 1] | 1 [1 to 1]
  gp70-TV1.GSKvacV1V2/293F (Month 36): number analyzed (Participants) | 25 | 26 | 6
  gp70-TV1.GSKvacV1V2/293F (Month 36) | 1 [1 to 130.5] | 7.625 [1 to 93.25] | 1 [1 to 1]

40. Secondary Outcome: Part B: Occurrence of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine in the Extension Study, at 6 Months After the Month 30 Vaccination
Description: as for outcome 13
Time Frame: Measured at Month 30 and 36
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
Participants
  Any gp120 (Month 30): number analyzed (Participants) | 26 | 28 | 7
  Any gp120 (Month 30) | 18 | 17 | 0
  Any gp120 (Month 36): number analyzed (Participants) | 26 | 27 | 6
  Any gp120 (Month 36) | 18 | 16 | 0
  1086 gp120 (Month 30): number analyzed (Participants) | 26 | 28 | 7
  1086 gp120 (Month 30) | 12 | 8 | 0
  1086 gp120 (Month 36): number analyzed (Participants) | 26 | 27 | 6
  1086 gp120 (Month 36) | 11 | 12 | 0
  TV1 gp120 (Month 30): number analyzed (Participants) | 26 | 28 | 7
  TV1 gp120 (Month 30) | 16 | 15 | 0
  TV1 gp120 (Month 36): number analyzed (Participants) | 26 | 27 | 6
  TV1 gp120 (Month 36) | 17 | 12 | 0
  ZM96 gp120 (Month 30): number analyzed (Participants) | 24 | 27 | 6
  ZM96 gp120 (Month 30) | 15 | 14 | 0
  ZM96 gp120 (Month 36): number analyzed (Participants) | 24 | 25 | 6
  ZM96 gp120 (Month 36) | 15 | 13 | 0

41. Secondary Outcome: Part B: Level of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine in the Extension Study, at 6 Months After the Month 30 Vaccination
Description: as for outcome 13
Time Frame: Measured at Month 30 and 36
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
Number analyzed (Participants) | 32 | 31 | 7
% CD4+ T-cells
  Any gp120 (Month 30): number analyzed (Participants) | 26 | 28 | 7
  Any gp120 (Month 30) | 0.128764915 [0.06016473 to 0.27276348] | 0.10384047 [0.066876795 to 0.13216669] | 0.00929931 [0.00092681 to 0.014916]
  Any gp120 (Month 36): number analyzed (Participants) | 26 | 27 | 6
  Any gp120 (Month 36) | 0.115994935 [0.05879524 to 0.23501344] | 0.09751639 [0.04296324 to 0.13914346] | 0.007663255 [0.00606286 to 0.01858776]
  1086 gp120 (Month 30): number analyzed (Participants) | 26 | 28 | 7
  1086 gp120 (Month 30) | 0.07396858 [0.02441189 to 0.12233446] | 0.05696544 [0.03144404 to 0.07578682] | 0.00878693 [-0.00320097 to 0.01448971]
  1086 gp120 (Month 36): number analyzed (Participants) | 26 | 27 | 6
  1086 gp120 (Month 36) | 0.064916705 [0.0324317 to 0.13007222] | 0.06119621 [0.0304561 to 0.09814416] | 0.001323895 [-0.00945559 to 0.01858776]
  TV1 gp120 (Month 30): number analyzed (Participants) | 26 | 28 | 7
  TV1 gp120 (Month 30) | 0.114625195 [0.05209329 to 0.20612288] | 0.077949675 [0.03458573 to 0.119078365] | -0.00139331 [-0.00836455 to 0.00929931]
  TV1 gp120 (Month 36): number analyzed (Participants) | 26 | 27 | 6
  TV1 gp120 (Month 36) | 0.106333215 [0.05700492 to 0.22142132] | 0.04974197 [0.03854645 to 0.11333829] | -0.00506502 [-0.01127566 to 0.00837665]
  ZM96 gp120 (Month 30): number analyzed (Participants) | 24 | 27 | 6
  ZM96 gp120 (Month 30) | 0.09879441 [0.041524935 to 0.2188063] | 0.08841848 [0.04422036 to 0.13041836] | -0.006057945 [-0.01286774 to 0.0063703]
  ZM96 gp120 (Month 36): number analyzed (Participants) | 24 | 25 | 6
  ZM96 gp120 (Month 36) | 0.104756745 [0.0461914 to 0.19649763] | 0.10113899 [0.01625771 to 0.1234859] | -0.001777015 [-0.01008356 to 0.00631053]

ADVERSE EVENTS:
Time Frame: Serious adverse events are collected throughout the study (months 0-18 for Part A, and months 30-36 for Part B). Non-serious adverse events are collected through 30 days after each vaccination (at months 0, 1, 3, 6, and 12 for Part A, and month 30 for Part B).
Arm/Group | Part A, Group 1: Vaccine | Part A, Group 2: Placebo | Part B, Group 1a: Vaccine | Part B, Group 1b: Vaccine/Placebo | Part B, Group 2: Placebo
All-Cause Mortality (participants affected / at risk) | 2/210 | 0/42 | 0/32 | 0/31 | 0/7
Serious Adverse Events (participants affected / at risk) | 7/210 | 0/42 | 0/32 | 0/31 | 0/7
Other Adverse Events (participants affected / at risk) | 147/210 | 34/42 | 15/32 | 18/31 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: Vaccine (N=210) | Part A, Group 2: Placebo (N=42) | Part B, Group 1a: Vaccine (N=32) | Part B, Group 1b: Vaccine/Placebo (N=31) | Part B, Group 2: Placebo (N=7)
Any Event in SOC (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Group 1: Vaccine (N=210) | Part A, Group 2: Placebo (N=42) | Part B, Group 1a: Vaccine (N=32) | Part B, Group 1b: Vaccine/Placebo (N=31) | Part B, Group 2: Placebo (N=7)
Any Event in SOC (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 20 (23) | 7 (10) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 22 (29) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 18 (21) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 81 (112) | 24 (27) | 10 (12) | 10 (10) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 0 (0)
Genitourinary tract gonococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 8 (9) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 32 (35) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urogenital trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 23 (26) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Buttock injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear canal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 48 (75) | 8 (11) | 1 (1) | 7 (7) | 1 (1)
Alanine aminotransferase increased (Investigations) | 19 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 22 (26) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 7 (9) | 0 (0) | 1 (1) | 6 (6) | 1 (1)
Blood pressure increased (Investigations) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (2) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urobilinogen urine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 14 (15) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 18 (21) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 14 (15) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature ejaculation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 19 (23) | 3 (4) | 2 (2) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 13 (14) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 14 (16) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Abnormal withdrawal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 13 (19) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT02404311/Prot_SAP_ICF_000.pdf